CLINICAL TRIAL: NCT02068313
Title: Phase II Study of Whole or Partial Parotid Sparing Intensity Modulated Radiotherapy in Patients With Head and Neck Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 3301
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Single cohort
  Interventions: Radiation: Toxicity and outcome measures of IMRT

INTERVENTIONS:
Radiation: Toxicity and outcome measures of IMRT

SUMMARY:
Phase II and III studies have demonstrated IMRT to be safe and standard practice for head and neck cancers treated with radiotherapy. This study will be an extension to an earlier, in-house, trial to allow continued recording of toxicities and outcomes in patients receiving IMRT for head and neck cancers. This study will allow us to examine radiobiological modelling for normal tissue complication probability and in particular, determining the dose threshold for parotid glands. Our primary objective is to assess the potential effectiveness of intensity-modulated radiotherapy (IMRT) in reducing xerostomia in head and neck cancer patients and determining threshold dose for whole parotid gland and superficial lobes of parotid glands

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell cancer or undifferentiated cancer of nasopharynx, oropharynx, larynx and hypopharynx and squamous cell carcinoma unknown primary.
* TNM Stage: T1-4, N0-3 M0
* Patients requiring primary or postoperative radiotherapy to the primary site and bilateral neck irradiation requiring IMRT
* Parotid sparing IMRT feasible (parotids clear of malignant disease)
* WHO Performance status 0-1 (Karnofsky >80)
* Aged 18 or older
* Induction chemotherapy and concomitant platinum based chemotherapy is permitted
* Concomitant cetuximab is permitted where platinum chemotherapy is contraindicated
* All patients must be suitable to attend regular follow-up and salivary flow measurements and be available for long term follow up.
* All patients must be able to complete self-assessed quality of life questionnaire
* Be able to provide written informed consent

Exclusion Criteria:

* Previous radiotherapy to the parotid gland/s
* Pre-existing salivary gland pathology interfering with saliva production
* Previous or concurrent illness which in the investigator's opinion which will interfere with either completion of therapy or follow up
* Brachytherapy is not allowed as part of the treatment
* Presence of lymphadenopathy adjacent to or involving both parotid glands making whole parotid sparing or superficial parotid sparing impossible
* Prophylactic use of amifostine or pilocarpine is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed squamous cell cancer or undifferentiated cancer of nasopharynx, oropharynx, larynx and hypopharynx and squamous cell carcinoma unknown primary referred for primary or postoperative radiotherapy to the primary site and bilateral neck irradiation requiring IMRT
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
To assess the potential effectiveness of intensity-modulated radiotherapy (IMRT) in reducing xerostomia in head and neck cancer patients and determining threshold dose for whole parotid gland and superficial lobes of parotid glands | 5 years

SECONDARY OUTCOMES:
To quantify acute and late toxicities of IMRT to provide data for radiobiological modelling (eg xerostomia, mucositis and dysphagia) | 5 years
Overall survival | 5 years
Disease free survival | 5 years
Loco-regional control | 5 years
General and specific QoL | 5 years
Xerostomia related QoL | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nutting, PhD, MD, FRCR, MRCP, MB BS, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Royal Marsden Hospital, Sutton, Surrey
  - The Royal Marsden Hospital, London